CLINICAL TRIAL: NCT01590589
Title: REGISTRY - an Observational Study of the European Huntington's Disease Network (EHDN)
Acronym: REGISTRY
Status: Completed | Type: Observational
Sponsor: European Huntington's Disease Network (Network)
Responsible Party: Sponsor
Other Study IDs: REGISTRY 3.0
Record Dates: First submitted 2012-03-22; First posted 2012-05-03 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Huntington Disease; Huntington's Disease
Keywords: Huntington Disease; European HD Network; Cohort; REGISTRY; EHDN
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — * DNA from whole blood
  * DNA
  * Lymphoblastoid cell lines
  * Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- REGISTRY participants: Individuals
  * with manifest HD
  * unaffected but known to carry the HD mutation
  * unaffected but at risk of carrying the HD mutation
  * from HD families known not to carry the HD mutation
  * from outside HD families acting as control research participants (e.g., spouses)

SUMMARY:
This is a multi-centre, multi-national, prospective, observational study of Huntington's disease (HD) with a control group of volunteers to:

* obtain natural history data on many HD mutation carriers and individuals who are part of an HD family
* relate phenotypical characteristics (genetic modifiers / wet and dry biomarkers)
* expedite identification and recruitment of participants for clinical trials
* develop and validate sensitive and reliable outcome measures for detecting onset and change over the natural course of premanifest and manifest HD which may also be potential outcome measures for use in future clinical trials and clinical care
* plan for future research studies

DETAILED DESCRIPTION:
REGISTRY integrates prospectively and systematically collected clinical research data (e.g. phenotypical clinical features, family history, demographical characteristics) with access to biological specimens (e.g. blood, urine) obtained from individuals with manifest HD, unaffected individuals known to carry the HD mutation or at risk of carrying the HD mutation, and control research participants (e.g. spouses, siblings or offspring of HD mutation carriers known not to carry the HD mutation).

REGISTRY is an open-ended study and eligible subjects are assessed at annual study visits on the phenotypical characteristics of HD regardless of whether they display clinical symptoms and signs of the disease and of individuals who are part of an HD family (irrespective of their mutation carrier status). At each study visit, general clinical, motor function, behavior, cognitive, Health Economics, Quality of Life assessments are administered. In addition, participants are given the option to consent to the donation of biosamples for the purposes of mutation (CAG repeat length) testing and for research to identify biological modifiers and markers of HD. Biological specimens and phenotypical data are made available to qualified scientists whose projects are reviewed and approved by the Scientific and Bioethical Advisory Committee (SBAC) of EHDN. Successful applicants agree to accept the EHDN policies surrounding the use of the data/materials provided and publication of results (see data sharing and publication policies of EHDN, attached). Research projects should aim to advance scientific knowledge towards establishing clinically effective treatments that delay onset and/or slow the progression of the disease.

ELIGIBILITY:
REGISTRY-HD participants include those who are willing to participate in regular (annual) evaluations conducted by the investigators and have a diagnosis of HD, are HD mutation carriers (but who do not meet criteria for a diagnosis of HD) or persons at risk for HD (first and second degree relatives of people affected by HD), are non-HD mutation carrier relatives. Spouses of participants may take part as REGISTRY-CONTROLS.

Inclusion Criteria:

The following individuals may be eligible to participate

* Individuals, confirmed HD mutation carrier
* Manifest HD, without mutation (CAG) testing
* HD family member at-risk, without CAG testing
* HD family member, non-HD mutation carrier
* REGISTRY-CONTROL participants: companion/individual without HD history
* REGISTRY-COMPANION (any of the above).

Exclusion Criteria:

* Participants who are unable to understand the study protocol or unable to give informed consent, and have no legal representative.
* Participants with choreic movement disorder other than HD. (EHDN provides a Registry-like tool to record findings in patients affected with choreatic movement disorders other than HD under the label "Neuroacanthocytosis"; www.euro-hd.net/html/na/registry).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with manifest HD, unaffected individuals known to carry the HD mutation or at risk of carrying the HD mutation, and control research participants (e.g., spouses, siblings or offspring of HD mutation carriers known not to carry the HD mutation)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2004-06; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Phenotypical characteristics of HD | 13 years
  The goal of the project is to collect longitudinal data on the phenotypical characteristics of HD gene mutation carriers.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Landwehrmeyer, Professor, Principal Investigator — University Hospital of Ulm / Dept. of Neurology
Locations (140):
- Austria (2):
  - Universitätsklinik für Psychiatrie, Neuropsychiatrische Ambulanz, Graz
  - Universitätsklinik Innsbruck, Neurologie, Innsbruck
- Belgium (3):
  - UCL-St Luc, Centre de génétique humaine, Brussels
  - Institute of Pathology and Genetics (IPG), Gosselies
  - Universitair Ziekenhuis Gasthuisberg, Dienst Neurologie, Leuven
- Czechia (2):
  - Fakultní nemocnice Olomouc, Neurologická klinika, Olomouc
  - Centrum extrapyramidových onemocnění, Neurologická klinika, 1. LFUK, Prague
- University Hospital of Copenhagen - Rigshospitalet, Dept. of Neurology, Copenhagen Ø, Denmark
- Finland (8):
  - The Family Federation of Finland Väestöliitto, Department of Medical Genetics, Helsinki
  - Helsinki University Hospital, Dept. of Neurology, HUS
  - Kuopio University Hospital, Neurology, Kuopio
  - Ålands Hälso- och Sjukvård, Långvårdsenheten, Mariehamn
  - Oulu University Hospital (OUH), Dept. of Neurology, Oulu
  - Suomen Terveystalo, Tampere
  - Turku University Hospital, Dept. of Neurology, Turku
  - The Finnish Parkinson Association, Suvituuli, Turku
- France (11):
  - CHU d'Amiens - Hôpital Nord, Service de Neurologie, Amiens
  - CHU d'Angers, Service de Neurologie Charcot, Angers
  - Hôpital Pellegrin, Service de Génétique Médicale (ESF 3e étage), Bordeaux
  - HU Clermont-Ferrand - Hôpital Gabriel Montpied, Service de Neurologie, Clermont-Ferrand
  - Hôpital Henri Mondor, Service de Neurologie, Créteil
  - Clinique Neurologique Hôpital Roger Salengro CHRU, Neurologie et Pathologie du Mouvement, Lille
  - CHU La Timone, Service de Neurologie (9e étage), Marseille
  - Hôpital La Pitié Salpétrière, Génétique & Inserm U679, Paris
  - CHU Rouen Charles Nicolle, Service de Neurologie, Rouen
  - Hôpital Civil, Service de Neurologie, Strasbourg
  - Hôpital Purpan, INSERM U825, Pôle Neurosciences, Toulouse
- Germany (17):
  - Universitätsklinikum Aachen, Neurologische Klinik, Aachen
  - Charité - Universitätsmedizin Berlin, Klinik und Poliklinik für Neurologie, Klinik für Psychiatrie und Psychotherapie, Berlin
  - Ruhruniversität Bochum, Neurologie, Bochum
  - Reha-Zentrum Dinslaken im Gesundheitszentrum Lang, Tagesklinik, Dinslaken
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Klinik und Poliklinik für Neurologie, Dresden
  - Universtität Erlangen, Abteilung für Molekulare Neurologie, Erlangen
  - Universitätsklinikum Freiburg, Neurologie, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Neurologische Abteilung, Hamburg
  - Neurologische Klinik mit Klinischer Neurophysiologie, Medizinische Hochschule Hannover, Hanover
  - Psychatrium Gruppe AöR, Haus 2/1, Heiligenhafen
  - Schwerpunktpraxis Huntington, Neurologie-Psychiatrie, Itzehoe
  - Praxis, Marburg
  - Universität Marburg, Neurologie, Marburg
  - Technische Universität München, Abteilung Neurologie, München
  - Universitätsklinikum Münster, Klinik und Poliklinik für Neurologie, Münster
  - Isar-Amper-Klinikum - Klinik Taufkirchen (Vils), Taufkirchen
  - University Hospital of Ulm, Dept. of Neurology, Ulm
- Italy (12):
  - University of Bari, Dept. of Neurological and Psychiatric Sciences, Bari
  - Università di Bologna, Dip. di Scienze Neurologiche - Clinica Neurologica, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Clinica Neurologica, Brescia
  - University of Florence, Dip. di Scienze Neurologiche e Psichiatriche, Florence
  - Università di Genova, Dept. of Neurosciences, Genova
  - Fondazione IRCCS Istituto Neruologico Carlo Besta, SOSD Genetics of Neurodegenerative and Metabolic Diseases, Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, I Neurologia, Milan
  - Università di Napoli Federico II, Dip. Scienze Neurologiche Edificio 17, Napoli
  - Azienda Ospedaliera Universitarie Pisana, Dip. di Neuroscienze - UO Neurologia, Pisa
  - IRCCS Neuromed, U.O. Neurogenetica, Pozzilli (IS)
  - Azienda Ospedaliera S. Andrea, UOC Neurologia e Centro Neurologico Terapie Sperimentali CENTERS, Rome
  - Università Cattolica del Sacro Cuore "A.Gemelli", Istituto di Neurologia / CNR, Istituto di Farmacologia Traslazionale, Rome
- Netherlands (4):
  - Medisch Spectrum Twente, Dept. of Neurology, Enschede
  - UMC Groningen, Neurology, Groningen
  - Leiden University Medical Centre (LUMC), Neurology K5-Q, Leiden
  - MUMC, Dept. Neurology, Maastricht
- Norway (4):
  - NKS Olaviken Alderpsykiatriske sykehus, Poliklinikk og Huntington Klinikk, Bergen
  - Rikshospitalet, Dept. of Medical Genetics, Oslo
  - Ulleval University Hospital, Medical Genetics, Oslo
  - St. Olavs Hospital HF, Neurology, Trondheim
- Poland (6):
  - Specialistic Hospital in Gdansk, Dept. of Neurology, Gdansk
  - Medical University of Silesia, Dept. of Neurology, Katowice
  - Krakowska Akademia Neurologii, Krakow
  - Poznan University of Medical Sciences, Dept. of Social Medicine, Poznan
  - Medical University of Warsaw, Dept. of Neurology, Warsaw
  - Institute of Psychiatry and Neurology, First Dept. of Neurology, Warsaw
- Portugal (7):
  - Hospital de Coimbra, Neurology Dept., Coimbra
  - Hospital dos Capuchos, Centro Hospitalar Lisboa Central, Neurology Dept., Lisbon
  - Hospital de Santa Maria, Centro de Estudos Egas Moniz, Neurology Dept., Lisbon
  - Hospital Fernando Fonseca, Neurology Dept., Lisbon
  - Hospital de São João, Neurology Dept., Porto
  - Hospital Geral de Santo António, Neurology Dept., Porto
  - Centro Hospitalar de Trás-os-Montes e Alto Douro, Neurology Dept., Vila Real
- Huntington's Disease Society of Russia, Moscow, Russia
- Spain (23):
  - Complejo Hospitalario Universitario de Albacete, Neurología, Albacete
  - Hospital Infanta Cristina, Neurología, Badajoz
  - Hospital Vall d'Hebrón, Neurología, 3ª planta, consultas externas, Barcelona
  - Hospital Clínic i Provincial, Neurología, Barcelona
  - Hospital Bellvitge, Neurología, Barcelona
  - Hospital General Yagüe, Neurology, Burgos
  - Hospital Puerta del Mar, Neurología, Cadiz
  - Centro Ramón y Cajal, Neurología, Madrid
  - Fundación Jiménez Díaz, Neurology, Madrid
  - Hospital Clínico de Madrid, Servicio de Neurología, Madrid
  - Hospital de Fuenlabrada, Neurology, Madrid
  - Hospital Virgen de la Arrixaca, Neurology, Murcia
  - Hospital Central de Oviedo, Neurología, Oviedo
  - Hospital Son Dureta, Neurology, Palma de Mallorca
  - Hospital Virgen del Camino, Medical Genetics, Pamplona
  - Hospital Donostia. Universidad del Pais Vasco, Neurociencias, San Sebastián
  - Hospital General de Segovia, Neurología, Segovia
  - Hospital Universitario Virgen del Rocío, Servicio de Neurología, Seville
  - Hospital Virgen Macarena, Neurología, Seville
  - Hospital Universitario Mutua de Terrassa, Neurologia - Investigación, Terrassa - Barcelona
  - Hospital Virgen de la Salud, Neurology, Toledo
  - Hospital La Fe, Consultas Externas de Neurología, Valencia
  - Hospital Clinico Universario, Department of Neurology, Zaragoza
- Sweden (6):
  - Sahlgren University Hospital, Dept. of Clinical Genetics, Gothenburg
  - Skåne Universitetssjukhus, Neurologiska kliniken, Lund
  - Neuroenheten Utsikten, Stockholm
  - Karolinska University Hospital - Huddinge Division, Neurology, Stockholm
  - Norrlands Universitet Sjukhus, Dept. of Neurology, Umeå
  - Uppsala University Hospital, Neurology, Uppsala
- Switzerland (3):
  - Neurologische Klinik des Inselspitals, Praxis, Bern
  - CHUV - Centre Hospitalier Universitaire Vaudois, Département de Neurologie, Lausanne
  - University Hospital Zurich, Dept. of Neurology, Zurich
- United Kingdom (30):
  - Clinical Genetics Centre, Ground Floor, Ashgrove House, Aberdeen
  - The Barberry Centre, Dept. of Psychiatry, Birmingham
  - Blandford Hospital, Blandford Forum
  - Frenchay Hospital, Neurology Dept., Bristol
  - Cambridge Centre for Brain Repair, Forvie Site, Cambridge
  - Cardiff University, Life Sciences Building, Cardiff
  - Ninewells Hospital and Medical School, Human Genetics Unit, Dundee
  - Molecular Medicine Centre, Western General Hospital, Dept. of Clinical Genetics, Edinburgh
  - Royal Devon and Exeter Foundation Trust Hospital, Department of Neurology, Exeter
  - Queen Margaret Hospital, Fife
  - Scottish Huntington Association, Units 105/106, Glasgow
  - Gloucestershire Royal Hospital, Neurology Dept., Gloucester
  - Chapel Allerton Hospital, Yorkshire Regional Genetics Service, Hull
  - Chapel Allerton Hospital, Leeds
  - Leicestershire Partnership NHS Trust, EMD South School, OSL house, Leicester
  - The Walton Centre for Neurology and Neurosurgery, Liverpool
  - Guy's Hospital, Dept. of Neurology, London
  - The Royal Hospital for Neuro-disability, Research and Development, London
  - St George's Hospital Medical School, South West Thames Regional Genetics Unit, London
  - National Hospital for Neurology and Neurosurgery, Dept. for Neurology, London
  - University of Manchester, Genetic Medicine, St. Mary's Hospital, Manchester
  - Institute of Human Genetics, International Centre for Life, Newcastle upon Tyne
  - Churchill Hospital, Dept. of Clinical Genetics, Oxford
  - Derriford Hospital, Dept. of Clinical Neuropsychology, Plymouth
  - Poole Hospital Foundation Trust, Brain Injury Service, Poole
  - Lancashire Teaching Hospitals NHS Foundation Trust, Neurosciences Directorate, Royal Preston Hospital, Preston
  - Sheffield Children's Hospital, Dept. of Clinical Genetics, Sheffield
  - Southampton General Hospital and University of Southampton, Neurology / Wellcome Trust Clinical Research Facility, Southampton
  - Bucknall Hospital, Neuropsychiatry Service, Stoke-on-Trent
  - Victoria Centre, Swindon

REFERENCES:
- [Result] Rickards H, De Souza J, van Walsem M, van Duijn E, Simpson SA, Squitieri F, Landwehrmeyer B; European Huntington's Disease Network. Factor analysis of behavioural symptoms in Huntington's disease. J Neurol Neurosurg Psychiatry. 2011 Apr;82(4):411-2. doi: 10.1136/jnnp.2009.181149. Epub 2010 Apr 14. PMID 20392980
- [Result] Orth M, Handley OJ, Schwenke C, Dunnett SB, Craufurd D, Ho AK, Wild E, Tabrizi SJ, Landwehrmeyer GB; Investigators of the European Huntington's Disease Network. Observing Huntington's Disease: the European Huntington's Disease Network's REGISTRY. PLoS Curr. 2010 Sep 28;2:RRN1184. doi: 10.1371/currents.RRN1184. PMID 20890398
- [Result] Orth M; European Huntington's Disease Network; Handley OJ, Schwenke C, Dunnett S, Wild EJ, Tabrizi SJ, Landwehrmeyer GB. Observing Huntington's disease: the European Huntington's Disease Network's REGISTRY. J Neurol Neurosurg Psychiatry. 2011 Dec;82(12):1409-12. doi: 10.1136/jnnp.2010.209668. Epub 2010 Nov 19. No abstract available. PMID 21097549
- [Result] Busse M, Al-Madfai DH, Kenkre J, Landwehrmeyer GB, Bentivoglio A, Rosser A; European Huntington's Disease Network. Utilisation of Healthcare and Associated Services in Huntington's disease: a data mining study. PLoS Curr. 2011 Jan 21;3:RRN1206. doi: 10.1371/currents.RRN1206. PMID 21304753
- [Result] Lopez-Sendon JL, Royuela A, Trigo P, Orth M, Lange H, Reilmann R, Keylock J, Rickards H, Piacentini S, Squitieri F, Landwehrmeyer B, Witjes-Ane MN, Jurgens CK, Roos RA, Abraira V, de Yebenes JG; European HD Network. What is the impact of education on Huntington's disease? Mov Disord. 2011 Jul;26(8):1489-95. doi: 10.1002/mds.23385. Epub 2011 Mar 22. PMID 21432905
- [Result] Ho AK, Hocaoglu MB; European Huntington's Disease Network Quality of Life Working Group. Impact of Huntington's across the entire disease spectrum: the phases and stages of disease from the patient perspective. Clin Genet. 2011 Sep;80(3):235-9. doi: 10.1111/j.1399-0004.2011.01748.x. Epub 2011 Aug 4. PMID 21736564
- [Result] Quarrell OW, Handley O, O'Donovan K, Dumoulin C, Ramos-Arroyo M, Biunno I, Bauer P, Kline M, Landwehrmeyer GB; European Huntington's Disease Network. Discrepancies in reporting the CAG repeat lengths for Huntington's disease. Eur J Hum Genet. 2012 Jan;20(1):20-6. doi: 10.1038/ejhg.2011.136. Epub 2011 Aug 3. PMID 21811303
- [Result] Saft C, Epplen JT, Wieczorek S, Landwehrmeyer GB, Roos RA, de Yebenes JG, Dose M, Tabrizi SJ, Craufurd D; REGISTRY Investigators of the European Huntington's Disease Network; Arning L. NMDA receptor gene variations as modifiers in Huntington disease: a replication study. PLoS Curr. 2011 Oct 4;3:RRN1247. doi: 10.1371/currents.RRN1247. PMID 21989477
- [Result] Rickards H, De Souza J, Crooks J, van Walsem MR, van Duijn E, Landwehrmeyer B, Squitieri F, Simpson SA; European Huntington's Disease Network. Discriminant analysis of Beck Depression Inventory and Hamilton Rating Scale for Depression in Huntington's disease. J Neuropsychiatry Clin Neurosci. 2011 Fall;23(4):399-402. doi: 10.1176/jnp.23.4.jnp399. PMID 22231310
- [Result] Lee JM, Ramos EM, Lee JH, Gillis T, Mysore JS, Hayden MR, Warby SC, Morrison P, Nance M, Ross CA, Margolis RL, Squitieri F, Orobello S, Di Donato S, Gomez-Tortosa E, Ayuso C, Suchowersky O, Trent RJ, McCusker E, Novelletto A, Frontali M, Jones R, Ashizawa T, Frank S, Saint-Hilaire MH, Hersch SM, Rosas HD, Lucente D, Harrison MB, Zanko A, Abramson RK, Marder K, Sequeiros J, Paulsen JS; PREDICT-HD study of the Huntington Study Group (HSG); Landwehrmeyer GB; REGISTRY study of the European Huntington's Disease Network; Myers RH; HD-MAPS Study Group; MacDonald ME, Gusella JF; COHORT study of the HSG. CAG repeat expansion in Huntington disease determines age at onset in a fully dominant fashion. Neurology. 2012 Mar 6;78(10):690-5. doi: 10.1212/WNL.0b013e318249f683. Epub 2012 Feb 8. PMID 22323755
- [Result] Henley SM, Ridgway GR, Scahill RI, Kloppel S, Tabrizi SJ, Fox NC, Kassubek J; EHDN Imaging Working Group. Pitfalls in the use of voxel-based morphometry as a biomarker: examples from huntington disease. AJNR Am J Neuroradiol. 2010 Apr;31(4):711-9. doi: 10.3174/ajnr.A1939. Epub 2009 Dec 24. PMID 20037137
- [Result] Aziz NA, Jurgens CK, Landwehrmeyer GB; EHDN Registry Study Group; van Roon-Mom WM, van Ommen GJ, Stijnen T, Roos RA. Normal and mutant HTT interact to affect clinical severity and progression in Huntington disease. Neurology. 2009 Oct 20;73(16):1280-5. doi: 10.1212/WNL.0b013e3181bd1121. Epub 2009 Sep 23. PMID 19776381
- [Derived] Stanislawska-Sachadyn A, Krzeminski M, Zielonka D, Krygier M, Zietkiewicz E, Slawek J, Limon J; REGISTRY investigators of the European Huntington's Disease Network (EHDN). Sex contribution to average age at onset of Huntington's disease depends on the number of (CAG)n repeats. Sci Rep. 2024 Jul 8;14(1):15729. doi: 10.1038/s41598-024-64105-5. PMID 38977715
- [Derived] Youssov K, Audureau E, Vandendriessche H, Morgado G, Layese R, Goizet C, Verny C, Bourhis ML, Bachoud-Levi AC. The burden of Huntington's disease: A prospective longitudinal study of patient/caregiver pairs. Parkinsonism Relat Disord. 2022 Oct;103:77-84. doi: 10.1016/j.parkreldis.2022.08.023. Epub 2022 Aug 24. PMID 36084356
- [Derived] McAllister B, Gusella JF, Landwehrmeyer GB, Lee JM, MacDonald ME, Orth M, Rosser AE, Williams NM, Holmans P, Jones L, Massey TH; REGISTRY Investigators of the European Huntington's Disease Network. Timing and Impact of Psychiatric, Cognitive, and Motor Abnormalities in Huntington Disease. Neurology. 2021 May 11;96(19):e2395-e2406. doi: 10.1212/WNL.0000000000011893. Epub 2021 Mar 25. PMID 33766994
- [Derived] Cubo E, Ramos-Arroyo MA, Martinez-Horta S, Martinez-Descalls A, Calvo S, Gil-Polo C; European HD Network. Clinical manifestations of intermediate allele carriers in Huntington disease. Neurology. 2016 Aug 9;87(6):571-8. doi: 10.1212/WNL.0000000000002944. Epub 2016 Jul 8. PMID 27402890
- See also: EHDN — http://www.euro-hd.net